CLINICAL TRIAL: NCT01565408
Title: Safety and Tolerability of NNC0114-0006 Following Multiple s.c. Dosing at Escalating Dose Levels in Subjects With Rheumatoid Arthritis
Brief Title: Safety and Tolerability of NNC0114-0006 at Increasing Dose Levels in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8828-3841; 2011-003037-33 (EudraCT Number); U1111-1122-4067 (Other: WHO)
Record Dates: First submitted 2012-03-21; First posted 2012-03-28 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Inflammation; Rheumatoid Arthritis
MeSH Terms: conditions — Inflammation; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NNC0114-0006 (Experimental)
  Interventions: Drug: NNC0114-0006
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: NNC0114-0006 — Multiple subcutaneous (s.c., under the skin) doses administered every second week for six weeks. The trial comprises dose escalation up to four dose levels. Progression to next dose will be based on safety evaluation.
  Arms: NNC0114-0006
Drug: placebo — Multiple subcutaneous (s.c., under the skin) doses administered every second week for six weeks.
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe. The aim of this dose-escalating trial is to assess the safety and tolerability of multiple doses of NNC0114-0006 in subjects with rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of RA, meeting the 2010 ACR-EULAR (American College of Rheumatology-European League Against Rheumatism) or the 1987 ACR classification criteria, made at least 4 months prior to trial drug administration
* Active RA, characterised by a DAS28-CRP equal to or above 4.5 and at least 5 tender and 5 swollen joints
* Methotrexate (MTX) treatment for at least 16 weeks (dose equal to or above 7.5 mg/week and equal to or below 25 mg/week) at a stable dose for at least 6 weeks prior to dosing
* Female subjects not pregnant and not nursing

Exclusion Criteria:

* Subjects with chronic inflammatory autoimmune disease other than RA
* Any active or ongoing chronic infectious disease requiring systemic anti-infectious treatment within 4 weeks prior to randomisation
* Body mass index (BMI) below 18.0 or above 35.0 kg/m^2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | From first administration of trial product (week 1) and up until week 27

SECONDARY OUTCOMES:
Change in serum levels of total IL-21 from first administration of trial product | Week 1, week 27
Change in disease activity score 28 calculated using C-reactive protein (DAS28-CRP) | From week 1 to week 9 (8 weeks after initiation of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (3):
- Novo Nordisk Investigational Site, Berlin, Germany
- Russia (2):
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Yaroslavl

REFERENCES:
- [Result] Wagner F, Skrumsager B, Fitilev S. Safety and tolerability of NNC0114-0006, an anti-IL-21 monoclonal antibody, at multiple s.c. dose levels in patients with rheumatoid arthritis. Arthritis and Rheumatology; 66 (10 (Supplement)): Abstract 1492
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com